CLINICAL TRIAL: NCT04359290
Title: Ruxolitinib for Treatment of Covid-19 Induced Lung Injury ARDS A Single-arm, Open-label, Proof of Concept Study
Brief Title: Ruxolitinib for Treatment of Covid-19 Induced Lung Injury ARDS
Acronym: RuXoCoil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KKS-278
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2020-11

CONDITIONS: ARDS, Human; COVID
Keywords: Covid-19; ARDS; Ruxolitinib; Janus kinase; JAK1; JAK2
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: Ruxolitinib will be administered p.o. or by gavage feeding starting with 2 x 10mg or 2 x 15mg bid dose at day 1 according to the investigator's decision and can be increased up to 2 x 15mg bid from day 2 to day 28 (max) (depending on platelet counts and renal function). Ruxolitinib will be administered in the morning and evening. Dosing will be adjusted according to toxicity and kidney function; open design, single arm.If the patient is discharged before day 28, the therapy will be discontinued for discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib treatment (Experimental): Ruxolitinib will be administered p.o. or by gavage feeding for max 28 days
  Interventions: Drug: Ruxolitinib administration

INTERVENTIONS:
Drug: Ruxolitinib administration — Ruxolitinib will be administered p.o. or by gavage feeding starting with 2 x 10mg or 2 x 15mg bid dose at day 1 according to the investigator's decision and can be increased up to 2 x 15mg bid from day 2 to day 28 (max) (depending on platelet counts and renal function). Ruxolitinib will be administered in the morning and evening. Dosing will be adjusted according to toxicity and kidney function.If the patient is discharged before day 28, the therapy will be discontinued for discharge.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ruxolitinib in the treatment of patients with COVID-19 severe pneumonia.

DETAILED DESCRIPTION:
This clinical trial is an open-label trial of ruxolitinib for the treatment of severe COVID-19 to assess its efficacy and safety.

Ruxolitinib (INCB018424 phosphate, INC424, ruxolitinib phosphate) is a well established, potent and selective inhibitor of Janus kinase (JAK)1 and JAK2, with modest to marked selectivity against tyrosine kinase (TYK)2 and JAK3, respectively. Ruxolitinib interferes with the signaling of a number of cytokines and growth factors that are important for hematopoiesis and immune function.

Ruxolitinib (JAKAVI®) is currently approved in the European Union (EU) for the treatment of disease-related splenomegaly or symptoms in adult patients with primary myelofibrosis (PMF) (also known as chronic idiopathic MF), post-polycythemia vera myelofibrosis (PPV-MF) or post-essential thrombocythemia myelofibrosis (PET-MF) and for the treatment of adult patients with PV who are resistant to or intolerant of hydroxyurea (HU). In the US, ruxolitinib has been approved in the treatment of steroid refractory graft versus host disease post allogeneic stem cell transplantation.

Because many patients with severe respiratory disease due to COVID-19 have features consistent with the cytokine release syndrome (CRS) and increased activation of the JAK/STAT pathway, it is postulated that ruxolitinib might have a useful role in treating these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female adult ≥18 years of age at time of enrollment.
2. has laboratory-confirmed SARS-CoV-2 infection as determined by PCR or other commercial or public health assay (result of the PCR is not necessary for inclusion, but has to approved latest within 48-72 hours after registration)
3. Willingness of men and women of childbearing potential to use highly effective contraceptive methods by abstinence or by using at least two contraceptive methods from the date of consent to the end of the study
4. severe lung disease as defined by following:

   1. Recent intubation
   2. Requirement of invasive ventilation moderate to severe pulmonary oxygen exchange disturbance as defined by (PaO2/FiO2) ≤ 200 mmHg at a PEEP ≥ 5mm H2O
   3. Serum LDH > 283 U/l
   4. Ferritin above normal value
   5. CT-scan: pulmonary infiltration compatible with Covid-19 disease
5. Patient or patient´s representative must provide written informed consent (and assent if applicable) before any study assessment is performed.

Exclusion Criteria:

1. Uncontrolled HIV infection
2. Active tuberculosis (result of positive tuberculosis infection is not necessary for exclusion, but has to approved later on during patient´s intervention)
3. Chronic kidney disease requiring dialysis
4. ALT/AST > 5 times the upper limit of normal.
5. Pregnancy or breast feeding.
6. Allergy to study medication
7. Simultaneous participation in another clinical trial with an experimental treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 28 days after registration into trial
  To determine the efficacy of ruxolitinib measured by overall survival

SECONDARY OUTCOMES:
Assessment of the duration of ventilation support | registration until 90 days after registration into trial
  Assessment of the duration of ventilation support
cytokine storm | registration until 90 days after registration into trial
  Assessment of the extent of cytokine storm reduction (IL-6, CRP, ferritin)
time on ICU | registration until 90 days after registration into trial
  To assess time on ICU
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | registration until 90 days after registration into trial
  In order to classify the severity of the AEs, number of participants with treatment-related adverse events will be assessed by the "Common Terminology Criteria for Adverse Events" (CTCAE) version 5.0
time frame for seroconversion under ruxolitinib treatment (SARS-Co-19- IgG) | registration until 90 days after registration into trial
  To assess the timeframe for seroconversion under ruxolitinib treatment (SARS-Co-19- IgG)
Rates of flow | Discharge from hospital (end of treatment)
  To asses the rates of flow (liter/minute), in order to detect possible amelioration of pulmonary function after Covid-19 infection
Gas exchange | Discharge from hospital (end of treatment)
  To asses gas exchange (partial pressure of oxygen and carbon dioxide), in order to detect possible amelioration of pulmonary function after Covid-19 infection
Forced expiratory volume in 1 second (FEV1) | Discharge from hospital (end of treatment)
  To assess forced expiratory volume in 1 second (liters), in order to detect possible possible amelioration of pulmonary function after Covid-19 infection
Forced vital capacity (FVC) | Discharge from hospital (end of treatment)
  To assess forced vital capacity (liters), in order to detect possible possible amelioration of pulmonary function after Covid-19 infection
Tiffeneau-Pinelli index | Discharge from hospital (end of treatment)
  To assess Tiffeneau-Pinelli index (FEV1/FVC ratio in %), in order to detect possible possible amelioration of pulmonary function after Covid-19 infection
Overall survival | 90 days after registration into trial
  To determine the efficacy of ruxolitinib measured by overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Neubauer, Prof Dr., Principal Investigator — Universitätsklinikum Giessen und Marburg (UKGM)
Locations (1):
- Andreas Neubauer, Marburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be provided after publication
Supporting Information: Study Protocol
Time Frame: 3 Months after publication
Access Criteria: Central server

REFERENCES:
- [Background] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Xia W, Shao J, Guo Y, Peng X, Li Z, Hu D. Clinical and CT features in pediatric patients with COVID-19 infection: Different points from adults. Pediatr Pulmonol. 2020 May;55(5):1169-1174. doi: 10.1002/ppul.24718. Epub 2020 Mar 5. PMID 32134205
- [Background] Wei M, Yuan J, Liu Y, Fu T, Yu X, Zhang ZJ. Novel Coronavirus Infection in Hospitalized Infants Under 1 Year of Age in China. JAMA. 2020 Apr 7;323(13):1313-1314. doi: 10.1001/jama.2020.2131. PMID 32058570
- [Background] [WHO] World Health Organization. Clinical management of severe acute respiratory infection when novel coronavirus (nCoV) infection is suspected [Resource on the internet]. 2020 [updated 13 March 2020; cited 24 March 2020]. Available from: https://www.who.int/publications-detail/clinical-management-of-severe-acute-respiratory-infection-when-novel-coronavirus-(ncov)-infection-is-suspected
- [Background] An Insight of comparison between COVID-19 (2019-nCoV disease) and SARS in pathology and pathogenesis. Author: Xiaolong Cai; Internet posting, of 27-Feb-2020 retrieved 24-Mar-2020. Cite as DOI: 10.31219/osf.io/hw34x
- [Background] Hermans MAW, Schrijver B, van Holten-Neelen CCPA, Gerth van Wijk R, van Hagen PM, van Daele PLA, Dik WA. The JAK1/JAK2- inhibitor ruxolitinib inhibits mast cell degranulation and cytokine release. Clin Exp Allergy. 2018 Nov;48(11):1412-1420. doi: 10.1111/cea.13217. Epub 2018 Aug 3. PMID 29939445
- [Background] Zhao J, Yu H, Liu Y, Gibson SA, Yan Z, Xu X, Gaggar A, Li PK, Li C, Wei S, Benveniste EN, Qin H. Protective effect of suppressing STAT3 activity in LPS-induced acute lung injury. Am J Physiol Lung Cell Mol Physiol. 2016 Nov 1;311(5):L868-L880. doi: 10.1152/ajplung.00281.2016. Epub 2016 Sep 16. PMID 27638904
- [Background] Coon TA, McKelvey AC, Lear T, Rajbhandari S, Dunn SR, Connelly W, Zhao JY, Han S, Liu Y, Weathington NM, McVerry BJ, Zhang Y, Chen BB. The proinflammatory role of HECTD2 in innate immunity and experimental lung injury. Sci Transl Med. 2015 Jul 8;7(295):295ra109. doi: 10.1126/scitranslmed.aab3881. PMID 26157031
- [Background] Ruxolitinib Prevents Cytokine Release Syndrome after CART Cell Therapy without Impairing the Anti-Tumor Effect in a Xenograft Model Saad S Kenderian, MD , Blood (2016) 128 (22): 652
- [Background] Calbet M, Ramis I, Calama E, Carreno C, Paris S, Maldonado M, Orellana A, Calaf E, Pauta M, De Alba J, Bach J, Miralpeix M. Novel Inhaled Pan-JAK Inhibitor, LAS194046, Reduces Allergen-Induced Airway Inflammation, Late Asthmatic Response, and pSTAT Activation in Brown Norway Rats. J Pharmacol Exp Ther. 2019 Aug;370(2):137-147. doi: 10.1124/jpet.119.256263. Epub 2019 May 13. PMID 31085698
- [Background] The definition and risks of Cytokine Release Syndrome-Like in 11 COVID-19-Infected Pneumonia critically ill patients: Disease Characteristics and Retrospective Analysis Wenjun Wang Jr. et al Internet posting of 27-Feb-2020 retrieved 24-Mar-2020 Cite as: https://doi.org/10.1101/2020.02.26.20026989
- [Background] Hoffmann J, Machado D, Terrier O, Pouzol S, Messaoudi M, Basualdo W, Espinola EE, Guillen RM, Rosa-Calatrava M, Picot V, Benet T, Endtz H, Russomando G, Paranhos-Baccala G. Viral and bacterial co-infection in severe pneumonia triggers innate immune responses and specifically enhances IP-10: a translational study. Sci Rep. 2016 Dec 6;6:38532. doi: 10.1038/srep38532. PMID 27922126
- [Derived] Neubauer A, Johow J, Mack E, Burchert A, Meyn D, Kadlubiec A, Torje I, Wulf H, Vogelmeier CF, Hoyer J, Skevaki C, Muellenbach RM, Keller C, Schade-Brittinger C, Rolfes C, Wiesmann T. The janus-kinase inhibitor ruxolitinib in SARS-CoV-2 induced acute respiratory distress syndrome (ARDS). Leukemia. 2021 Oct;35(10):2917-2923. doi: 10.1038/s41375-021-01374-3. Epub 2021 Aug 12. PMID 34385593